CLINICAL TRIAL: NCT07320989
Title: Impact of Chewing Gum on Bowel Preparation Quality and Tolerance in Patients Undergoing Colonoscopy With Split-Dose Bowel Preparation: A Randomized Controlled Trial
Brief Title: Impact of Chewing Gum on Bowel Preparation in Patients Undergoing Colonoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Ekta Gupta, Professor of Gastroenterology, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00115658
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer Screening
Keywords: Colonoscopy; Bowel Preparation; Chewing gum; Split-Dose PEG; Boston Bowel Preparation Scale; Patient Tolerance; Randomized Controlled Trial
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: This is a prospective, endoscopist-blinded, randomized controlled trial with 1:1 allocation to gum chewing (intervention) or control (no gum) during bowel preparation. Participants in both groups undergo standard split-dose bowel prep with either high-volume (4L PEG) or low-volume (2L PEG + adjunct) regimens, prescribed per clinical indication.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chewing Gum During Bowel Preparation (2L PEG-ELP) (Experimental): Participants randomized to the experimental arm will chew one piece of sugar-free gum for approximately 15-20 minutes, 30 minutes before starting the first dose of split-dose bowel preparation and again 30 minutes after the second dose. The gum is sugar-free and non-medicated. Participants will be instructed not to swallow the gum and to discontinue chewing if they experience discomfort.
  All participants will receive standard bowel preparation (either 4L PEG or 2L PEG + ascorbate, prescribed according to clinical indication).
  The endoscopist performing the colonoscopy will remain blinded to group assignment.
  Interventions: Behavioral: Chewing Sugar-Free Gum During Bowel Preparation; Other: Standard Bowel Prep (2L PEG-ELP)
- Standard Bowel Preparation 4L (No Gum) (Active Comparator): Participants in the control arm will undergo standard split-dose bowel preparation (4L PEG) according to clinical indication, without chewing gum before or after the preparation.
  Endoscopists will be blinded to participant group assignment.
  Interventions: Other: Standard Bowel Prep
- Chewing Gum During 4L Bowel Preparation (Experimental): Arm Description: Participants randomized to the experimental arm will chew one piece of sugar-free gum for approximately 15-20 minutes, 30 minutes before starting the first dose of split-dose bowel preparation and again 30 minutes after the second dose. The gum is sugar-free and non-medicated. Participants will be instructed not to swallow the gum and to discontinue chewing if they experience discomfort. All participants will receive standard bowel preparation (either 4L PEG or 2L PEG + ascorbate, prescribed according to clinical indication). The endoscopist performing the colonoscopy will remain blinded to group assignment.
  Interventions: Behavioral: Chewing Sugar-Free Gum During Bowel Preparation; Other: Standard Bowel Prep
- Standard Bowel Preparation 2L PEG-ELP (No Gum) (Active Comparator): Arm Description: Participants in the control arm will undergo standard split-dose bowel preparation (2L PEG + ascorbate) according to clinical indication, without chewing gum before or after the preparation. Endoscopists will be blinded to participant group assignment.
  Interventions: Other: Standard Bowel Prep (2L PEG-ELP)

INTERVENTIONS:
Behavioral: Chewing Sugar-Free Gum During Bowel Preparation — Participants randomized to the intervention arm will chew one piece of sugar-free gum for approximately 15-20 minutes, 30 minutes before the first dose of split-dose polyethylene glycol (PEG) bowel preparation and again 30 minutes after completing the second dose.
  The gum-chewing activity is intended to improve tolerance and satisfaction with the bowel preparation process through cephalic-vagal stimulation ("sham feeding") without altering the underlying cleansing regimen.
  Other Names: Chewing gum
  Arms: Chewing Gum During 4L Bowel Preparation; Chewing Gum During Bowel Preparation (2L PEG-ELP)
Other: Standard Bowel Prep (2L PEG-ELP) — Participants in this comparator arm will follow standard split-dose polyethylene glycol (PEG) bowel preparation (either 4L PEG or 2L PEG + ascorbate, prescribed per clinical indication) without gum chewing before or after the preparation.
  This represents the standard-of-care approach currently used for colonoscopy preparation at the study site.
  Arms: Chewing Gum During Bowel Preparation (2L PEG-ELP); Standard Bowel Preparation 2L PEG-ELP (No Gum)
Other: Standard Bowel Prep — Participants in this comparator arm will follow standard split-dose polyethylene glycol (PEG) bowel preparation (4L PEG, prescribed per clinical indication) without gum chewing before or after the preparation. This represents the standard-of-care approach currently used for colonoscopy preparation at the study site.
  Arms: Chewing Gum During 4L Bowel Preparation; Standard Bowel Preparation 4L (No Gum)

SUMMARY:
Colorectal cancer is the second leading cause of cancer deaths that could be prevented in the United States. Colonoscopy is the best test for finding and removing polyps before they turn into cancer. However, many people are hesitant to have a colonoscopy because of the bowel preparation. The preparation can be difficult to tolerate, with patients often struggling to finish it due to the taste, volume, or side effects like nausea and bloating. This can lead to incomplete procedures or discourage people from getting screened at all.

Chewing sugar-free gum is a simple, low-cost, and safe intervention that may make the preparation process easier. One study from China found that chewing gum did not change the quality of bowel cleansing, but patients reported that they were more satisfied with the process. No U.S.-based studies have tested this strategy, and no prior research has looked at whether gum chewing has different effects in people using high-volume versus low-volume prep solutions.

The investigators will randomize 160 participants to the stated intervention or control using computer-generated 1:1 randomization. Upon completing the study, the investigators will analyze the data.

By studying gum chewing during bowel preparation, the investigators hope to find out whether this small change can make bowel prep more tolerable and encourage more patients to complete their colonoscopy. If successful, this approach could help more people get screened, leading to earlier detection and prevention of colorectal cancer in the community.

DETAILED DESCRIPTION:
Background and Rationale Colorectal cancer (CRC) remains the second leading cause of preventable cancer-related death in the United States, with approximately 150,000 new cases and 50,000 deaths annually. Colonoscopy is the gold-standard screening modality for CRC because it allows both detection and removal of precancerous lesions within the same procedure. However, the success of colonoscopy depends heavily on adequate bowel cleansing. Suboptimal bowel preparation can lead to missed lesions, prolonged procedure times, and incomplete examinations, ultimately reducing screening effectiveness.

One of the most common barriers to successful colonoscopy completion is the patient's difficulty tolerating bowel preparation. Poor tolerance-due to the taste, volume burden, nausea, bloating, or abdominal discomfort associated with polyethylene glycol (PEG)-based solutions-can result in incomplete ingestion of the prep solution and inadequate cleansing. These experiences often discourage patients from future screening, contributing to low adherence to recommended screening guidelines, particularly among underserved populations.

Chewing gum has been proposed as a simple and low-cost adjunct that could improve tolerance to bowel preparation. The act of chewing gum stimulates cephalic-vagal pathways through "sham feeding," promoting gastrointestinal motility without adding calories or affecting electrolyte balance. In postoperative and perioperative gastrointestinal contexts, gum chewing has been shown to accelerate recovery of bowel function. A few small randomized controlled trials (RCTs) have evaluated gum chewing during bowel preparation, with mixed results. The largest study, conducted in China (n=300), found no improvement in cleansing quality but higher patient satisfaction. Other smaller studies in Turkey and elsewhere suggested improved tolerability and, in some regimens, enhanced cleansing scores.

To date, no prospective, randomized, endoscopist-blinded studies in the United States have investigated the impact of gum chewing on bowel preparation quality and patient experience using modern split-dose PEG regimens. Furthermore, no study has systematically compared outcomes between high-volume (4L PEG) and low-volume (2L PEG + ascorbate) preparations-two regimens that differ in both cost and tolerability and are commonly prescribed based on insurance coverage and comorbidities.

This study aims to address this gap by testing whether a benign, widely available behavioral intervention-chewing sugar-free gum before and after split-dose bowel preparation-can improve tolerance, satisfaction, and potentially the quality of bowel cleansing.

Study Objectives

Primary Objective:

To determine whether chewing sugar-free gum before and after split-dose bowel preparation improves bowel cleansing quality, measured by the Boston Bowel Preparation Scale (BBPS), compared with standard bowel preparation alone.

Secondary Objectives:

* To evaluate whether gum chewing improves patient tolerance to bowel preparation (nausea, bloating, cramping, discomfort).
* To assess overall satisfaction with the preparation process and willingness to repeat the prep in the future.
* To compare prep completion rates between the gum-chewing and control groups.
* To evaluate cecal intubation rates, procedure metrics (withdrawal time, total duration), and adenoma detection rates (ADR).
* To explore differences in outcomes between high-volume (4L PEG) and low-volume (2L PEG + ascorbate) subgroups.

Study Design This is a single-center, prospective, randomized, endoscopist-blinded controlled trial conducted at the University of Maryland Medical System (UMMC Midtown Campus) Outpatient Endoscopy Suite in Towson, Maryland.

Participants will be randomized in a 1:1 ratio to either:

Experimental Arm: Standard split-dose PEG bowel preparation + chewing sugar-free gum before and after the prep, or Active Comparator Arm: Standard split-dose PEG bowel preparation without gum chewing.

Both arms will undergo standard colonoscopy for clinical indications (screening, surveillance, or diagnostic).

Randomization will be performed using a computer-generated randomization sequence with equal allocation (n = 80 per arm, total n = 160). Endoscopists assessing bowel cleansing will remain blinded to group assignment.

Study Procedures

Recruitment and Consent:

Eligible patients will be identified during routine clinic visits when their colonoscopy is scheduled. The study will be explained by the principal investigator or trained research personnel in a private setting, and informed consent will be obtained.

Study Activities:

* Randomization (1:1) will occur after consent.
* Participants will follow their assigned bowel prep instructions.
* Nursing staff will record tolerance and satisfaction scores during pre-procedure intake.
* The blinded endoscopist will assess bowel cleansing using the Boston Bowel Preparation Scale (BBPS).

Additional data (prep completion, cecal intubation, procedure metrics, and ADR) will be abstracted from the electronic medical record.

Duration per Participant:

Each participant's involvement lasts approximately 24 hours-the time required to complete bowel preparation and the colonoscopy procedure. There is no post-procedure follow-up required for study purposes.

Total Study Duration:

The overall study is expected to take approximately two months, including start-up, enrollment, and analysis phases.

Sample Size and Statistical Analysis

Sample Size Calculation:

Assuming a moderate effect size (Cohen's d = 0.40) for improvement in tolerance/satisfaction, with a one-sided α = 0.05 and 80% power, approximately 78 participants per arm would be required. To accommodate potential dropouts and missing data, the investigators plan to enroll 160 participants total (80 per arm).

Analysis Plan:

Primary analysis: Comparison of mean total BBPS scores between the gum and control arms using a two-sample t-test or nonparametric equivalent (Wilcoxon rank-sum).

Secondary analyses:

* Chi-square or Fisher's exact tests for categorical variables (adequate vs inadequate cleansing, ADR, completion rates).
* Multivariable regression models to adjust for confounders (age, sex, BMI, prep type, comorbidities).
* Subgroup analyses comparing high-volume vs low-volume prep regimens.
* A p-value < 0.05 will be considered statistically significant.
* All analyses will be performed using de-identified data in a secure research environment (SRE).

Risks and Safety Considerations Chewing sugar-free gum is a low-risk activity. Potential risks include mild jaw discomfort, accidental swallowing of gum, or rarely choking. Participants will be instructed to chew only when seated and alert, to discard the gum after use, and to report any discomfort.

The bowel preparation carries standard, well-known risks such as nausea, bloating, cramps, or vomiting. Severe adverse events (e.g., dehydration, electrolyte imbalance, allergic reaction to PEG) are rare and will be managed per institutional protocols. Participants have access to clinical staff and an on-call physician for any adverse effects.

Loss of confidentiality is a minor risk; all identifying information will be stored separately from study data using password-protected, HIPAA-compliant systems.

Potential Benefits Participants may experience improved comfort or satisfaction during bowel preparation, although direct benefit cannot be guaranteed. The study findings may provide important information to improve the tolerability of colonoscopy preparation, enhance patient adherence, and ultimately support more effective colorectal cancer prevention strategies.

Data Management and Confidentiality Data will be abstracted from the electronic medical record (EPIC) and entered into an encrypted, password-protected Excel database within the Secure Research Environment (SRE). Identifiers such as name, date of birth, and medical record number will be used only for linkage and stored separately from analytic data. Each participant will be assigned a unique study ID. Access to data will be limited to authorized study personnel.

Research data will not be reused for other projects without IRB approval. De-identified aggregate results will be presented at scientific meetings and published in peer-reviewed journals.

Monitoring Plan Given the minimal-risk nature of the behavioral intervention, a formal data safety monitoring board (DSMB) is not required. The Principal Investigator will review all reported adverse events and protocol deviations, and any unanticipated problems will be reported promptly to the institutional IRB.

Ethical Considerations The study will be conducted in accordance with the ethical principles of the Declaration of Helsinki and the U.S. Common Rule (45 CFR 46). Informed consent will be obtained from all participants prior to enrollment. Participation is voluntary, and refusal or withdrawal will not affect clinical care.

Dissemination Plan Participants may opt to receive a lay summary of the results after study completion. Individual participant-level data will not be shared outside the research team.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years
* Scheduled for elective outpatient colonoscopy
* Able to provide informed consent

Exclusion Criteria:

* Prior major abdominal surgery (excluding appendectomy or cholecystectomy)
* Pregnancy
* Cognitive impairment
* Ward of the state
* Known allergy to PEG or gum components
* Current use of GI prokinetics
* Known temporomandibular joint (TMJ) disorder or difficulty chewing/swallowing

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bowel cleansing quality (BBPS total score) | Day of colonoscopy (intra-procedure assessment, immediately prior to withdrawal).
  Boston Bowel Preparation Scale (0-9; sum of right, transverse, left colon segment scores) assessed by the blinded endoscopist. Higher scores indicate better cleansing.

SECONDARY OUTCOMES:
Patient tolerance | Day of colonoscopy (pre-procedure)
  Global tolerance/symptom score (Likert or VAS) for nausea, bloating, cramps, and overall ease of prep recorded during routine pre-procedure nursing intake.
Patient satisfaction | Day of colonoscopy (pre-procedure)
  Single-item satisfaction rating (Likert) with the bowel preparation process, recorded by nursing staff.
Prep completion rate | Day of colonoscopy (pre-procedure)
  Proportion completing 100% of prescribed split-dose regimen vs partial/unknown, per intake documentation.
Willingness to repeat | Day of colonoscopy (pre-procedure)
  Willingness to repeat the same bowel prep in the future (yes/no or Likert).
Segmental Boston Bowel Preparation Scale (BPPS) Scores | Day of colonoscopy (intra-procedure)
  Right, transverse, and left colon BBPS segment scores.
  Boston Bowel Preparation Scale (0-9; sum of right, transverse, left colon segment scores) assessed by the blinded endoscopist. Higher scores indicate better cleansing.
Cecal intubation rate | Day of colonoscopy (intra-procedure)
  Successful cecal intubation (yes/no) per standard endoscopy report.
Adenoma detection rate (ADR) | Day of colonoscopy to 2 weeks post-procedure (to allow routine pathology posting)
  Proportion of colonoscopies with ≥1 histologically confirmed adenoma (if pathology recorded as part of usual care).
Procedure metrics | Day of colonoscopy
  Withdrawal time and total procedure duration (minutes).
Adverse events | Day of colonoscopy
  Immediate procedure-day AEs (e.g., gum-related issues reported at intake; standard colonoscopy AEs captured in recovery notes).

CONTACTS AND LOCATIONS:
Locations (1):
- UMMC Midtown - Outpatient Endoscopy Center, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Given the small, single-center RCT focused on workflow-embedded outcomes and minimal-risk behavioral exposure, the investigators do not plan to share de-identified IPD outside the study team. Aggregate results will be disseminated via presentations and peer-reviewed publication.

REFERENCES:
- [Result] Johnson DA, Barkun AN, Cohen LB, Dominitz JA, Kaltenbach T, Martel M, Robertson DJ, Boland CR, Giardello FM, Lieberman DA, Levin TR, Rex DK. Optimizing adequacy of bowel cleansing for colonoscopy: recommendations from the U.S. multi-society task force on colorectal cancer. Gastrointest Endosc. 2014 Oct;80(4):543-562. doi: 10.1016/j.gie.2014.08.002. No abstract available. PMID 25220509
- [Result] Gao C, Zou D, Wang W, Li Y, Han J, Su D, Qi X. Effect of chewing gum combined with WeChat-enhanced instruction on bowel preparation in constipated patients: a randomized-controlled trial. Gastroenterol Rep (Oxf). 2025 Apr 28;13:goaf034. doi: 10.1093/gastro/goaf034. eCollection 2025. PMID 40297539
- [Result] Guo T, et al. Chewing gum improves tolerance but not quality of bowel preparation: a systematic review and meta-analysis. World J Gastrointest Endosc. 2024;16(6):321-333.
- [Result] Atalay R, et al. Gum chewing improves bowel preparation quality for colonoscopy: a randomized trial. Turk J Gastroenterol. 2019;30(9):801-807.
- [Result] Zhang S, et al. Effect of chewing gum on bowel preparation before colonoscopy: a randomized controlled trial. Dis Colon Rectum. 2019;62(7):874-881.